CLINICAL TRIAL: NCT06854458
Title: The Multicenter Stress Cardiac Magnetic Resonance Quantitative Perfusion Imaging in the United States (SPINS2) Study
Brief Title: The Multicenter Stress Cardiac Magnetic Resonance Quantitative Perfusion Imaging in the United States Study
Acronym: SPINS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Raymond Y. Kwong, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024P003457
Record Dates: First submitted 2025-02-24; First posted 2025-03-03 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Heart Disease (IHD); Cardiac Magnetic Resonance Imaging; Myocardial Blood Flow
Keywords: Myocardial Blood Flow; Cardiac Magnetic Resonance; Quantitative perfusion; Cardiovascular Outcomes
MeSH Terms: conditions — Myocardial Ischemia | interventions — gadobutrol; Vasodilator Agents; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Myocardial Blood Flow Evaluation (Active Comparator): Qualitative stress cardiac magnetic resonance imaging only.
  Interventions: Diagnostic Test: Qualitative Myocardial Blood Flow Evaluation; Drug: Gadavist; Drug: Vasodilator; Diagnostic Test: Blood draw for the laboratory assessment
- New Myocardial Blood Flow Evaluation (Experimental): Quantitative + Qualitative stress cardiac magnetic resonance imaging.
  Interventions: Diagnostic Test: Quantitative Myocardial Blood Flow Evaluation; Drug: Gadavist; Drug: Vasodilator; Diagnostic Test: Blood draw for the laboratory assessment

INTERVENTIONS:
Diagnostic Test: Quantitative Myocardial Blood Flow Evaluation — The perfusion sequence will produce on-the-fly additional quantitative perfusion maps with segmental myocardial blood flow values.
  Other Names: New Myocardial Blood Flow Evaluation
  Arms: New Myocardial Blood Flow Evaluation
Diagnostic Test: Qualitative Myocardial Blood Flow Evaluation — The perfusion sequence will not produce additional quantitative perfusion maps.
  Other Names: Standard Myocardial Blood Flow Evaluation
  Arms: Standard Myocardial Blood Flow Evaluation
Drug: Gadavist — Participants will receive Gadavist 0.05 mmol/kg dose for each stress and rest perfusion imaging (total dose of 0.1 mmol/kg).
  Other Names: Gadobutrol
Drug: Vasodilator — All participants will receive vasodilator (regadenoson or adenosine depending on local site practice).
  Other Names: stress vasodilator
Diagnostic Test: Blood draw for the laboratory assessment — A single (7-10 ml tube) whole blood sample will be collected from each patient for processing of blood biomarkers.

SUMMARY:
This research aims to investigate whether symptoms of chest pain or shortness of breath among the study population are arising due to a heart problem, particularly any reduction of blood flow to the heart muscle from blockages in the coronary blood vessels or inflammation of the heart using cardiac magnetic resonance imaging that measures the amount of blood flow during a stress state meant to simulate vigorous exercise. At present, doctors use standard magnetic resonance imaging pictures of blood flow patterns to treat heart disease. The investigators want to study if detailed blood flow measurements, in addition to the standard blood flow pattern, could diagnose heart disease more accurately and allow more doctors to understand the severity of heart disease. Early research has demonstrated that detailed blood flow measurements may be more accurate in diagnosing heart disease in some patients, but doctors need more information to know how to use these measurements.

DETAILED DESCRIPTION:
In this proposal of the Multicenter Stress Cardiac Magnetic Resonance Quantitative Perfusion Imaging in the United States (SPINS2) study, the investigators seek to assess the prognostic utility of myocardial blood flow and flow reserve by quantitative stress cardiac magnetic resonance imaging compared to patients with normal quantitative perfusion indices. The investigators hypothesize that patients with abnormal myocardial blood flow and flow reserve will have higher adverse cardiac events, incremental to demographic risks and qualitative perfusion, and they should be considered for invasive workup or early institution of goal-directed medical therapies. In addition, the investigators hypothesize that quantitative perfusion by cardiac magnetic resonance imaging will characterize the myocardial extent and severity of multivessel disease and the participants' risk of adverse cardiac outcomes.

Patients with chest pain syndromes and suspected ischemic heart disease who meet both inclusion and exclusion criteria will be prospectively recruited among 20 sites across the United States over the course of 1.5 years. Participants will receive standardized quantitative stress cardiac magnetic resonance imaging protocol with Gadavist (Bayer, Germany) 0.05 mmol/kg dose for each stress and rest perfusion imaging (total dose of 0.1 mmol/kg) as per Food and Drug Administration (FDA)-approved indication. All participants will receive vasodilator stress with regadenoson or adenosine depending on local site practice. A single (7-10 ml tube) whole blood sample will be collected from each patient for processing of blood biomarkers.

All participants will have demographics and imaging characteristics recorded at baseline visits. Follow-up will occur via email or telephone at 3 months, 12 months, and 24 months from baseline. At each follow-up visit, medications, treatment, and adverse events will be recorded. In addition, all available electronic patient records will be reviewed in detail to capture all follow-up data which will be entered into an outline database using clearly defined data definitions. Participants will be followed for a total of 2 years from baseline cardiac magnetic resonance imaging study.

ELIGIBILITY:
Inclusion Criteria:

1. male or female at age 35-85 years,
2. presence of either of the following sign/symptom that led to a referral to stress cardiac magnetic resonance imaging:

   1. chest pain or anginal equivalent, or
   2. abnormal electrocardiogram with a suspicion of coronary artery disease
3. Intermediate or high risk of significant coronary disease based on at least 1 of the following conditions:

   a) patient age > 45 for male, 50 for female b) Diabetes, hypertension, or hypercholesterolemia: by either history or medical treatment c) family history of premature coronary disease: first degree relative at age <= 55 male and <=65 female d) history of smoking of > 10 packed-years e) post-menopausal state >5 years f) any chronic inflammatory conditions d) Body mass index > 30 e) Any medical documentation of coronary or peripheral artery disease

Exclusion Criteria:

1. Acute myocardial infarction within the past 30 days prior to cardiac magnetic resonance imaging
2. Confirmed diagnosis of any significant non-coronary cardiac conditions below:

   1. any severe-grade valvular heart disease,
   2. left ventricular ejection fraction <40% from any known non-coronary causes,
   3. infiltrative cardiomyopathy,
   4. hypertrophic cardiomyopathy,
   5. pericardial disease with significant constriction, or
3. active pregnancy,
4. any competing conditions leading to an expected survival of < 2 years
5. contraindication to vasodilator (regadenoson or adenosine)
6. metallic device or object that poses an magnetic resonance imaging safety hazard
7. metallic device with a high likelihood of non-diagnostic cardiac magnetic resonance images

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Primary composite outcome of major cardiovascular adverse events (MACE) | From cardiac magnetic resonance imaging to the end of follow-up in 24 months
  Composite MACE includes cardiovascular death, non-fatal acute myocardial infarction, stroke, resuscitated cardiac arrest, unnecessary invasive coronary angiography, and any cardiac hospitalization. Unnecessary invasive coronary angiography is defined as any invasive coronary angiography performed within 6 months after study enrollment, which reviews no obstructive coronary disease and no revascularization performed.

SECONDARY OUTCOMES:
Procedure-related complications | From cardiac magnetic resonance imaging to the end of follow-up in 24 months
  Serious complications from a coronary procedure (e.g., procedure-related myocardial infarction, stroke/Transient Ischemic Attack, major periprocedural bleeding, 50% reduction of estimated glomerular filtration rate (eGFR), or anaphylactic reaction).
Cost outcomes for Comparative Cost-effectiveness | From cardiac magnetic resonance imaging to the end of follow-up in 24 months
  Costs of performing coronary artery disease-related tests or procedures during the follow-up period, namely invasive coronary angiography; coronary revascularization procedure or surgery; any noninvasive stress imaging, stress electrocardiogram, or coronary computed tomography angiography imaging. Costs of performing these tests or procedures will be determined by national averaged Medicare cost of reimbursement adjusted across the years for rate of inflation.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pepine CJ, Anderson RD, Sharaf BL, Reis SE, Smith KM, Handberg EM, Johnson BD, Sopko G, Bairey Merz CN. Coronary microvascular reactivity to adenosine predicts adverse outcome in women evaluated for suspected ischemia results from the National Heart, Lung and Blood Institute WISE (Women's Ischemia Syndrome Evaluation) study. J Am Coll Cardiol. 2010 Jun 22;55(25):2825-32. doi: 10.1016/j.jacc.2010.01.054. PMID 20579539
- [Background] Patel MR, Peterson ED, Dai D, Brennan JM, Redberg RF, Anderson HV, Brindis RG, Douglas PS. Low diagnostic yield of elective coronary angiography. N Engl J Med. 2010 Mar 11;362(10):886-95. doi: 10.1056/NEJMoa0907272. PMID 20220183
- [Background] Sammut EC, Villa ADM, Di Giovine G, Dancy L, Bosio F, Gibbs T, Jeyabraba S, Schwenke S, Williams SE, Marber M, Alfakih K, Ismail TF, Razavi R, Chiribiri A. Prognostic Value of Quantitative Stress Perfusion Cardiac Magnetic Resonance. JACC Cardiovasc Imaging. 2018 May;11(5):686-694. doi: 10.1016/j.jcmg.2017.07.022. Epub 2017 Nov 15. PMID 29153572
- [Background] Kotecha T, Chacko L, Chehab O, O'Reilly N, Martinez-Naharro A, Lazari J, Knott KD, Brown J, Knight D, Muthurangu V, Hawkins P, Plein S, Moon JC, Xue H, Kellman P, Rakhit R, Patel N, Fontana M. Assessment of Multivessel Coronary Artery Disease Using Cardiovascular Magnetic Resonance Pixelwise Quantitative Perfusion Mapping. JACC Cardiovasc Imaging. 2020 Dec;13(12):2546-2557. doi: 10.1016/j.jcmg.2020.06.041. Epub 2020 Oct 1. PMID 33011115
- [Background] Patel AR, Kramer CM. Role of Cardiac Magnetic Resonance in the Diagnosis and Prognosis of Nonischemic Cardiomyopathy. JACC Cardiovasc Imaging. 2017 Oct;10(10 Pt A):1180-1193. doi: 10.1016/j.jcmg.2017.08.005. PMID 28982571
- [Background] Rozanski A, Gransar H, Hayes SW, Friedman JD, Hachamovitch R, Berman DS. Comparison of long-term mortality risk following normal exercise vs adenosine myocardial perfusion SPECT. J Nucl Cardiol. 2010 Dec;17(6):999-1008. doi: 10.1007/s12350-010-9300-9. Epub 2010 Nov 13. PMID 21076898
- [Background] Arai AE, Schulz-Menger J, Shah DJ, Han Y, Bandettini WP, Abraham A, Woodard PK, Selvanayagam JB, Hamilton-Craig C, Tan RS, Carr J, Teo L, Kramer CM, Wintersperger BJ, Harisinghani MG, Flamm SD, Friedrich MG, Klem I, Raman SV, Haverstock D, Liu Z, Brueggenwerth G, Santiuste M, Berman DS, Pennell DJ. Stress Perfusion Cardiac Magnetic Resonance vs SPECT Imaging for Detection of Coronary Artery Disease. J Am Coll Cardiol. 2023 Nov 7;82(19):1828-1838. doi: 10.1016/j.jacc.2023.08.046. PMID 37914512
- [Background] Nayfeh M, Ahmed AI, Saad JM, Alahdab F, Al-Mallah M. The Role of Cardiac PET in Diagnosis and Prognosis of Ischemic Heart Disease: Optimal Modality Across Different Patient Populations. Curr Atheroscler Rep. 2023 Jul;25(7):351-357. doi: 10.1007/s11883-023-01107-0. Epub 2023 May 10. PMID 37162723